CLINICAL TRIAL: NCT03685084
Title: Phase I, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of AAI101 Administered Intravenously Alone or in Combination With Piperacillin or Cefepime to Healthy Adult Subjects
Brief Title: Investigation of AAI101 Safety, Tolerability & PK in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allecra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: AT-101
Record Dates: First submitted 2018-09-19; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Healthy
MeSH Terms: interventions — enmetazobactam; Sodium Chloride; Monobactams

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.9% saline infusion (Placebo Comparator): Saline 0.9% infusion
  Interventions: Drug: AAI101 i.v.; Drug: Saline 0.9% infusion
- AAI101 i.v. (Experimental): 600 mg, 1g, 2g, 4g, 1g q6h, 2g q6h.
  Drug-Drug Interaction:
  Sequence 1 = piperacillin 4 g i.v. - AAI101 2 g i.v. - AAI101 2 g + piperacillin 4 g i.v. - cefepime 2 g i.v. - AAI101 2 g + cefepime 2 g i.v.
  Sequence 2 = cefepime 2 g i.v. - piperacillin 4 g i.v. - AAI101 2 g + cefepime 2 g i.v. - AAI101 2 g i.v. - AAI101 2 g + piperacillin 4 g i.v.
  Interventions: Drug: AAI101 i.v.; Drug: Saline 0.9% infusion
- Piperacillin i.v. (Experimental): Piperacillin 3 g
  Interventions: Drug: Piperacillin i.v.
- Cefepime i.v. (Experimental): Cefepime 1 g
  Interventions: Drug: Cefepime i.v.

INTERVENTIONS:
Drug: AAI101 i.v. — 600 mg, 1 g, 2 g, 4 g, 1 g (every 6h), 2 g (every 6h)
  Other Names: AAI101
  Arms: 0.9% saline infusion; AAI101 i.v.
Drug: Saline 0.9% infusion — Vehicle infusion
  Other Names: Vehicle
  Arms: 0.9% saline infusion; AAI101 i.v.
Drug: Piperacillin i.v. — piperacillin 3 g i.v.
  Other Names: Beta-lactam antibiotic
  Arms: Piperacillin i.v.
Drug: Cefepime i.v. — cefepime 1 g i.v.
  Other Names: Beta-lactam antibiotic
  Arms: Cefepime i.v.

SUMMARY:
* To assess the safety and tolerability of single and multiple ascending intravenous doses of AAI101 (SAD & MAD) in healthy male subjects.
* To assess the safety and tolerability of single and multiple ascending intravenous doses of AAI101 in combination with fixed intravenous doses of piperacillin or cefepime in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers aged between 18 and 45 years (inclusive) at screening.
* Body mass index (BMI) of 18.0 to 30.0 Kg/m2 (inclusive) at screening.
* Healthy as determined by the investigator on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12 lead ECG readings (all results were to be within normal range or considered non-clinically significant by the investigator).
* Non-smoker or smoker of fewer than 10 cigarettes per day as determined by medical history. Had to be able to abstain from smoking during the inpatient stay.
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.

Main Exclusion Criteria:

* Any significant cardiovascular (e.g., hypertension), hepatic, renal, respiratory (e.g., childhood asthma), gastrointestinal, endocrine (e.g., diabetes, dyslipidemia), immunologic, hematological, neurologic, or psychiatric disease.
* Acute disease state (e.g., nausea, vomiting, fever, diarrhea) within 7 days before study Day 1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects
Enrollment: 56 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-01-13 (Actual); Study Completion 2014-01-13 (Actual)

PRIMARY OUTCOMES:
Safety Profile - Number of Subjects With at Least one Adverse Event | Throughout the period that subjects receive study drug up to 5 days following discontinuation of study treatment
  Safety will be evaluated from reported signs and symptoms and clinical laboratory tests

SECONDARY OUTCOMES:
AAI101 maximum plasma concentration (Cmax) | Up to 24 hours post-dose
  Cmax will be compared before and after administration of AAI101 either alone or in the presence of cefepime or piperacillin
AAI101 Clast | Up to 24 hours post-dose
  Clast will be compared before and after administration of AAI101 either alone or in the presence of cefepime or piperacillin
AAI101 AUC(0-t) - AUC(0-8) | Up to 24 hours post-dose
  AAI101 Urea Under the Curve will be compared before and after administration of AAI101 either alone or in the presence of cefepime or piperacillin
AAI101 half life (t1/2) | Up to 24 hours post-dose
  AAI101 t1/2 plasma pharmacokinetic parameter will be compared for AAI101 alone or in the presence of cefepime or piperacillin

IPD SHARING:
Plan to Share IPD: No